CLINICAL TRIAL: NCT03434483
Title: Microbiome, Inflammation and Genetics as a Target for Precision Medicine in AThERosclerosis
Brief Title: The Microbiome as a Target for Precision Medicine in Atherosclerosis
Acronym: MIGATER
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Fundación para la Investigación Biomédica del Hospital Gregorio Maranon (Other)
Responsible Party: Principal Investigator, Javier Bermejo Thomas, MD PhD Cardiology Department HGUGM, Hospital General Universitario Gregorio Marañon
Other Study IDs: FIBHGM-MIGATER; PIE 16/00055 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2018-01-08; First posted 2018-02-15 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Acute Coronary Syndrome; Atherosclerosis
Keywords: Microbiota; Immunity; Genetics; Atherosclerosis
MeSH Terms: conditions — Acute Coronary Syndrome; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Feces, blood, salive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute Coronary Syndrome: Patients with an episode of acute coronary syndrome. Clinical evaluation 1 year. Gene variants in atherosclerosis. Microbiota analysis. Immunological analysis.
  Interventions: Genetic: Gene variants in atherosclerosis; Other: Microbiota analysis; Other: Immunological analysis; Other: Clinical evaluation
- ACS-Angiographic substudy: Patients included in the Acute Coronary Syndrome group with clinical indication for revascularization.
  Clinical evaluation. Assessment of the atherosclerotic plaque in a moderate lession at baseline and 1-year .
  Gene variants in atherosclerosis. Microbiota analysis. Immunological analysis
  Interventions: Procedure: Assessment of the atherosclerotic plaque in a moderate lession.; Genetic: Gene variants in atherosclerosis; Other: Microbiota analysis; Other: Immunological analysis; Other: Clinical evaluation
- Chronic coronary atherosclerosis: Patients with chronic atherosclerosis. Gene variants in atherosclerosis. Microbiota analysis. Immunological analysis.
  Interventions: Genetic: Gene variants in atherosclerosis; Other: Microbiota analysis; Other: Immunological analysis; Other: Clinical evaluation

INTERVENTIONS:
Procedure: Assessment of the atherosclerotic plaque in a moderate lession. — In patients who have been successfully revascularized the artery responsible for AMI and also present an intermediate lesion (40-80%) in another coronary territory, the clinical care protocol of the Cardiology Service stipulates the need for a physiological assessment with guidance of pressure (FFR).
  The thickness of the fibrous cap shall be measured using optical coherence tomography.
  In addition to the FFR measurement, a complete physiological assessment with a Doppler-pressure guide. This will allow the procedure to be performed without additional risk to the patient. The physiological study will include the analysis of endothelium-dependent vascular function and endothelium-independent vascular function.
  Other Names: Coronary blood collection
  Groups: ACS-Angiographic substudy
Genetic: Gene variants in atherosclerosis — From the blood samples of the patients, the total DNA will be extracted and the main functional variants identified in the literature will be genotyped
Other: Microbiota analysis — From the samples of blood, feces, oral cavity and blood, the DNA of the microbiota will be extracted using specific extraction kits and the microbiome will be analyzed through the study of 16S ribosomal RNA amplicons.
Other: Immunological analysis — A study of immunological cell populations and cytokines will be carried out from fresh blood samples using antibody panels and flow cytometry
Other: Clinical evaluation — Clinical evaluation including hemostasis and biochemical studies and questionaries for diet and exercice registration

SUMMARY:
Cardiovascular diseases are the main cause of death in industrialized countries. Among them, atherosclerosis has the highest prevalence and constitutes a common pathological pathway responsible for the majority of cases of chronic ischemic heart disease, acute myocardial infarction, heart failure and cerebrovascular disease. Classic studies have confirmed well-established etiopathogenic factors of atherosclerosis based on genetic and immunological components and environmental modifying agents such as diet and exercise. But in addition, recent experimental studies have shown that dysbiosis (alteration of the microbiota) may be an additional factor that participates in the onset and progression of atherosclerosis. The objective of this study is to identify the potential interactions between changes in the microbiota, changes in the immune status, the clinical evolution and the instability and progression of atherosclerosis.

DETAILED DESCRIPTION:
The study will prospectively study two groups of patients : 1) patients with acute coronary syndrome and 2) age and sex matched patients with chronic stable documented atherosclerosis.

Immune cell populations and immune-related metabolites will be characterized, the genetic profile of the main known functional variants will be determined, and the oral, gastrointestinal, and blood microbiota will be compared in both groups in a transversal observational design.

In addition, 1-year clinical follow-up will be performed and correlation with the evolution of the microbiota and immune response in a longitudinal design will be conducted.

Besides, an angiographic substudy, for those patients included in the study but that require revascularization of culprit artery according to clinical indication, will be 1 year follow-up and functional assessment and intravascular imaging and the degree of remodelling of the atherosclerotic plaque will be correlated with the evolution of the microbiota and immune response in a longitudinal design.

ELIGIBILITY:
Inclusion Criteria Acute coronary syndrome group:

* Diagnosis of acute coronary syndrome
* Signature of informed consent for the study (Annex I).

Exclusion Criteria Acute coronary syndrome group:

* Previous Ejection fraction of VI less than 30%.
* History of heart failure
* Systemic inflammatory diseases
* In treatment with corticosteroids or immunomodulators
* In treatment with antibiotics during the last month

Aditional Inclusion Criteria for angiographic substudy group:

* Clinical indication of coronary angiography in the acute phase (in the first 72 hours after its hospital diagnosis).
* At least one non-causal coronary lesion in a coronary segment with reference diameter> 2 mm, stenosis between 40-80%, and TIMI 3 flow in this vessel (angiographic criteria, only confirmed after performing coronary angiography)
* Signature of informed consent for the substudy (Annex II).

Aditional Exclusion Criteria for angiographic substudy group:

* Renal insufficiency with creatinine clearance less than 30 ml / h
* Hepatic insufficiency: patients with cirrhosis in Child B or C stages will be excluded.

Inclusion Criteria Chronic atherosclerosis group:

* Angiographic diagnosis, using catheterization or computed tomography of coronary atherosclerotic disease.
* Clinical situation of stable chronic ischemic heart disease.
* Signature of informed consent for the study (Annex III).

Exclusion Criteria Chronic atherosclerosis group:

* Previous Ejection fraction of VI less than 30%.
* History of heart failure
* Systemic inflammatory diseases
* In treatment with corticosteroids or immunomodulators
* In treatment with antibiotics during the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute coronary syndrome candidates for the study will be all patients with an episode of acute coronary syndrome wwho enter the Gregorio Marañón General University Hospital who meet all of the inclusion criteria and none of the exclusion criteria.
  Chronic atherosclerosis candidates for the study will be all patients with chronic atherosclerosis under follow-up in the General University Hospital Gregorio Marañón that meet all the following inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in clinical evaluation at 12 months | Inclusion, 1 week, 1 month, 3 months, 6 months and 12 months
  Cardiac events register including hemostasis and biochemical determinations
Change from baseline in fibrous cap thickness at 12 months | Inclusion and 12 months
  Angiographic substudy-Change from baseline in the thickness of the fibrous cap (μm) of an atherosclerotic plaque in the nonculprit vessel as measured using optical coherence tomography

SECONDARY OUTCOMES:
Endothelial dysfunction | Inclusion and 12 months
  Angiographic substudy-Micro and macrovascular endothelial function measured using a Doppler pressure guidewire
Intestinal microbiota composition changes 16S | Inclusion, 1 week, 1 month, 3 months, 6 months and 12 months
  Changes from baseline in intestinal microbiota will be analysed using the 16S rRNA target gene sequencing approach at 1 week, 1 month, 3 months, 6 months and 12 months
Intestinal microbiota composition changes metagenome | Inclusion, 1 week, 1 month, 3 months, 6 months and 12 months
  Changes from baseline in intestinal microbiota will be analysed using the metagenome sequencing approach at 1 week, 1 month, 3 months, 6 months and 12 months
Blood microbiota composition changes 16S | Inclusion, 1 week, 1 month, 3 months, 6 months and 12 months
  Changes from baseline in blood microbiota will be analysed using the 16S rRNA target gene sequencing approach at 1 week, 1 month, 3 months, 6 months and 12 months
Blood microbiota composition changes metagenome | Inclusion, 1 week, 1 month, 3 months, 6 months and 12 months
  Changes from baseline in blood microbiota will be analysed using the metagenome sequencing approach at 1 week, 1 month, 3 months, 6 months and 12 months
Oral microbiota composition changes 16S | Inclusion, 1 week, 1 month, 3 months, 6 months and 12 months
  Changes from baseline in oral microbiota will be analysed using the 16S rRNA target gene sequencing approach at 1 week, 1 month, 3 months, 6 months and 12 months
Oral microbiota composition changes metagenome | Inclusion, 1 week, 1 month, 3 months, 6 months and 12 months
  Changes from baseline in oral microbiota will be analysed using the genome sequencing approach at 1 week, 1 month, 3 months, 6 months and 12 months
Adaptive immune system status changes | Inclusion, 1 week, 1 month, 3 months, 6 months and 12 months
  Changes from baseline of adaptive immune cell lineages will be assessed dynamically using high performance cytometry at 1 week, 1 month, 3 months, 6 months and 12 months
Innate immune system status changes | Inclusion, 1 week, 1 month, 3 months, 6 months and 12 months
  Changes from baseline of innate immune cell lineages will be assessed dynamically using high performance cytometry at 1 week, 1 month, 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Fernández-Aviles, Prof, MD, Study Director — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital General Universitario Gregorio Maranon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] I Fernandez-Avila A, Gutierrez-Ibanes E, Martin de Miguel I, Sanz-Ruiz R, Gabaldon A, Fernandez-Aviles F, Gomez-Lara J, Fernandez-Castillo M, Vazquez-Cuesta S, Martinez-Legazpi P, Lozano-Garcia N, Blazquez-Lopez E, Yotti R, Lopez-Cade I, Reigadas E, Munoz P, Elizaga J, Correa R, Bermejo J. One-year longitudinal changes of peripheral CD4+ T-lymphocyte counts, gut microbiome, and plaque vulnerability after an acute coronary syndrome. Int J Cardiol Heart Vasc. 2024 Jun 4;53:101438. doi: 10.1016/j.ijcha.2024.101438. eCollection 2024 Aug. PMID 38912228